CLINICAL TRIAL: NCT00591539
Title: Carotid Artery Disease in Long-Term Survivors of Childhood Cancer
Brief Title: Carotid Artery Disease in Childhood Cancer Survivors
Status: Terminated | Type: Observational
Why Stopped: Slow Accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2006-0487
Record Dates: First submitted 2007-12-28; First posted 2008-01-11 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Pediatric Cancers
Keywords: Carotid Artery Disease; Intima-Media Thickening; Carotid Ultrasound; Pediatric Cancer Survivors; Cancer Survivors; Head or Neck Cancer; Radiation Therapy
MeSH Terms: conditions — Carotid Artery Diseases; Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Carotid Ultrasound: Carotid Ultrasound: Irradiated and non-irradiated sides of the neck in long-term survivors of pediatric cancers who received unilateral radiation therapy involving the carotid artery as part of their treatment
  Interventions: Procedure: Carotid Ultrasound

INTERVENTIONS:
Procedure: Carotid Ultrasound — Bilateral carotid ultrasound measurements: A test that uses sound waves to look at the blood vessels in the neck.

SUMMARY:
The goal of this clinical research study is to find out if long-term survivors of childhood head or neck cancer, who received radiation therapy as part of the overall treatment plan, are at increased risk of thickening or blockage of the carotid arteries (the major blood vessels in the neck).

Researchers also want to find out if other medical conditions, such as high blood sugar, high blood cholesterol, or history of tobacco use may contribute to the thickening or blockage of the carotid arteries.

DETAILED DESCRIPTION:
Some research shows that survivors of adult head or neck cancer, who received radiation therapy, are at increased risk for thickening or blockage of the carotid arteries, which may increase the risk for other medical conditions, such as stroke. Researchers want to learn about the possible risks of thickening or blockage of the carotid arteries in survivors of childhood head or neck cancer.

If you agree to take part in this study, researchers will see if there are any possible effects (thickening or blockage) of radiation therapy on your carotid arteries. This will be done by examining the test results from routine testing (mentioned below) that is normally done for your standard long-term follow-up care of the disease. These routine tests would be performed even if you were not in this research study.

During your long-term follow-up clinic appointment, you will have a physical exam and an ultrasound test (performed at the Cardiology Clinic) of the carotid arteries. A carotid ultrasound is a test that uses sound waves to look at the blood vessels in the neck. Blood will be drawn (about 2-3 teaspoons) for laboratory tests, including blood sugar level, blood cholesterol level, blood triglyceride level, thyroid hormone level, and blood levels of certain proteins (C-reactive protein and brain natriuretic peptide).

If any of the tests show any thickening or blockage of the carotid arteries or other medical problems, such as high blood sugar, your study doctor will discuss the test results, treatment options, and/or a follow-up plan with you.

This is an investigational study. Up to 60 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have been less than 21 years of age at time of initial diagnosis.
2. Patients treated at M.D. Anderson Cancer Center for any malignancy (including primary CNS tumors) that required unilateral radiation therapy to the head and neck area and involving the ipsilateral carotid artery as part of the overall treatment plan.
3. Patients must be at least 5 years status post completion of therapy.
4. Must be English speaking, or able to consent through an approved medical language translator.
5. A written informed consent from the patient and/or the patient's legally authorized guardian must be obtained from all patients.

Exclusion Criteria:

1. Leukemia patients receiving craniospinal irradiation
2. Non-English speaking subjects for which no appropriate medical translator is available
3. Patients who received head/neck radiation involving both carotid arteries will not be eligible.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Long-term survivors of pediatric cancers who received radiation therapy to the neck as part of their treatment at M.D. Anderson Cancer Center.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2007-12; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Patients with Carotid intima-media thickening (IMT) | Carotid ultrasound testing and laboratory examinations performed at time of routinely scheduled yearly appointment.

SECONDARY OUTCOMES:
Patients with Carotid artery stenosis (CAS) | Carotid ultrasound testing and laboratory examinations performed at time of routinely scheduled yearly appointment.

CONTACTS AND LOCATIONS:
Overall Officials: Winston Huh, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org